CLINICAL TRIAL: NCT05542394
Title: Determination of Pharmacokinetics of Different Curcuminoids Preparations: Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Collaborators: Nutritional Fundamentals for Health (Unknown)
Responsible Party: Principal Investigator, Shatha Hammad, Assistant Professor, Assistant Professor, University of Jordan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 10-2022/13342
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Plasma Levels of Different Curcuminoids Preparations
Keywords: Curcumin H2O, Tumeric, piperine
MeSH Terms: interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Curcumin H2O SAP (Experimental): Water soluble version of turmeric extract standardized to 10% curcuminoids will be administered orally (1 dose)
  Interventions: Dietary Supplement: Curcumin
- Tumeric with piperine SAP (Active Comparator): Turmeric extract standardized to 95% curcuminoids in combination with 5 mg of piperine per capsule will be administered orally (1 dose)
  Interventions: Dietary Supplement: Curcumin
- Tumeric without piperine (Placebo Comparator): Turmeric extract standardized to 95% curcuminoids without piperine will be administered orally (1 dose)
  Interventions: Dietary Supplement: Curcumin

INTERVENTIONS:
Dietary Supplement: Curcumin — water soluble version of turmeric extract standardized to 10% curcuminoids
  .
  Other Names: NFH

SUMMARY:
This pilot study aims to investigate the pharmacokinetics of a novel curcuminoid preparation with suggested high bioavailability due to its solubility in water, compared to two standard hydrophobic formulations. The findings of this study will help the health care providers and community to select suitable formulation.

DETAILED DESCRIPTION:
This pilot study is the first phase that must be followed, in the second phase, by longer clinical trials to support the findings and investigate the role of the novel preparation on health.The second phase will include an assessment of the effectiveness of several doses of curcumin preparation on health as well as an evaluation of the tolerance and possible adverse effects. The latter could not be evaluated at this stage of a single dose.

ELIGIBILITY:
Inclusion Criteria:

Male and female Apparently healthy adults

Exclusion Criteria:

Postmenopausal women Smokers Overweight Chronic diseases

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Blood concentration of bisdemethoxycurcumin | [Time Frame: Change during 8 hours]
  plasma bisdemethoxycurcumin levels using LC MS/MS
Blood concentration of desmethoxycurcumin | [Time Frame: Change during 8 hours]
  plasma desmethoxycurcumin levels using LC MS/MS
Blood concentration of piperine-curcuminoids | [Time Frame: Change during 8 hours]
  plasma piperine-curcuminoids levels using LC MS/MS
Blood concentration of hexahydrocurcumin | [Time Frame: Change during 8 hours]
  plasma hexahydrocurcumin levels using LC MS/MS
Blood concentration of curcumin diethyl disuccinate | [Time Frame: Change during 8 hours]
  plasma curcumin diethyl disuccinate levels using LC MS/MS
Blood concentration of tetrahydrocurcumin | [Time Frame: Change during 8 hours]
  plasma tetrahydrocurcumin levels using LC MS/MS
Blood concentration of curcumin | [Time Frame: Change during 8 hours]
  plasma curcumin levels using LC MS/MS

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sahebkar A, Henrotin Y. Analgesic Efficacy and Safety of Curcuminoids in Clinical Practice: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Pain Med. 2016 Jun;17(6):1192-202. doi: 10.1093/pm/pnv024. Epub 2015 Dec 14. PMID 26814259
- [Background] Schiborr C, Kocher A, Behnam D, Jandasek J, Toelstede S, Frank J. The oral bioavailability of curcumin from micronized powder and liquid micelles is significantly increased in healthy humans and differs between sexes. Mol Nutr Food Res. 2014 Mar;58(3):516-27. doi: 10.1002/mnfr.201300724. Epub 2014 Jan 9. PMID 24402825
- [Background] Kocher A, Bohnert L, Schiborr C, Frank J. Highly bioavailable micellar curcuminoids accumulate in blood, are safe and do not reduce blood lipids and inflammation markers in moderately hyperlipidemic individuals. Mol Nutr Food Res. 2016 Jul;60(7):1555-63. doi: 10.1002/mnfr.201501034. Epub 2016 May 23. PMID 26909743
- [Background] Fanca-Berthon P, Tenon M, Bouter-Banon SL, Manfre A, Maudet C, Dion A, Chevallier H, Laval J, van Breemen RB. Pharmacokinetics of a Single Dose of Turmeric Curcuminoids Depends on Formulation: Results of a Human Crossover Study. J Nutr. 2021 Jul 1;151(7):1802-1816. doi: 10.1093/jn/nxab087. PMID 33877323
- [Background] Kocher A, Schiborr C, Behnam D, Frank J: The oral bioavailability of curcuminoids in healthy humans is markedly enhanced by micellar solubilisation but not further improved by simultaneous ingestion of sesamin, ferulic acid, naringenin and xanthohumol.Journal of functional foods 2015, 14:183-191.
- [Background] Baum L, Cheung SK, Mok VC, Lam LC, Leung VP, Hui E, Ng CC, Chow M, Ho PC, Lam S, Woo J, Chiu HF, Goggins W, Zee B, Wong A, Mok H, Cheng WK, Fong C, Lee JS, Chan MH, Szeto SS, Lui VW, Tsoh J, Kwok TC, Chan IH, Lam CW. Curcumin effects on blood lipid profile in a 6-month human study. Pharmacol Res. 2007 Dec;56(6):509-14. doi: 10.1016/j.phrs.2007.09.013. Epub 2007 Sep 18. PMID 17951067
- [Background] Carroll RE, Benya RV, Turgeon DK, Vareed S, Neuman M, Rodriguez L, Kakarala M, Carpenter PM, McLaren C, Meyskens FL Jr, Brenner DE. Phase IIa clinical trial of curcumin for the prevention of colorectal neoplasia. Cancer Prev Res (Phila). 2011 Mar;4(3):354-64. doi: 10.1158/1940-6207.CAPR-10-0098. PMID 21372035
- [Background] Dhillon N, Aggarwal BB, Newman RA, Wolff RA, Kunnumakkara AB, Abbruzzese JL, Ng CS, Badmaev V, Kurzrock R. Phase II trial of curcumin in patients with advanced pancreatic cancer. Clin Cancer Res. 2008 Jul 15;14(14):4491-9. doi: 10.1158/1078-0432.CCR-08-0024. PMID 18628464